CLINICAL TRIAL: NCT03480841
Title: Enhancing Communication Between Children in EI and Their Depressed Mothers
Brief Title: Using the LENA System in Early Intervention - b
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-2105b
Record Dates: First submitted 2018-03-22; First posted 2018-03-29 (Actual); Results first posted 2019-12-06 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LENA with Feedback (Experimental): Mothers who will run the Language ENhancement Assessment/intervention system with their young children, and will receive initial feedback from researchers on LENA output and how to enhance the language the home language environment.
  Interventions: Behavioral: Language ENhancement Assessment/intervention system

INTERVENTIONS:
Behavioral: Language ENhancement Assessment/intervention system — The LENA with Feedback intervention will involve mothers running the Language ENhancement Assessment/intervention system, an audiorecorder language pedometer that records adult speech centered on the child, child vocalizations, and parent-child reciprocal turn-taking conversations. Researchers will provide an initial feedback session to mothers, which will include reviewing the LENA visual output from the previous recording and how mothers can access the output on their own for future recordings. Mothers will independently use the LENA system and access the output on their own.

SUMMARY:
This project will determine whether an intervention to enhance communication between infants and toddlers with developmental disabilities and their depressed mothers can be integrated into federally-funded Early Intervention (EI) services. Participants will be mothers with depressive symptoms whose children are receiving EI services, along with their EI service providers.

The investigators will conduct a small feasibility trial using the Language ENhancement Assessment/intervention system (LENA), a technology-supported language monitoring system, with 10 mothers and one of their child's EI service providers. The LENA uses an infant or toddler garment with an integrated audiotape system that records adult speech centered on the child, child vocalizations, and reciprocal parent-child turn-taking conversations. The LENA software produces visual feedback that a mother can use to focus her language interactions with her child. They study will follow participants in the LENA with feedback intervention over 6 weeks: 5 weeks of LENA data collection (with mothers running the system 1 day/week for 16 consecutive hours). The investigators will analyze data from measures on LENA communication data (adult word count, child vocalizations and conversational turn-taking), and measures of child language, maternal depressive symptoms, and child disability profiles.

DETAILED DESCRIPTION:
Early Intervention (EI) services are provided to infants and toddlers with documented developmental delays in all 50 states and US territories. EI improves long-term infant-toddler adaptation and lowers the cost of care if parents use the services. However, depressive symptoms can reduce mothers' ability to provide the daily child development-promoting activities recommended by EI, increasing the child's risk for communication and behavioral problems. Indeed, repeated studies have shown that depressive symptoms reduce mothers' consistent use of developmentally sensitive, child-centered speech which, in turn, lead to negative child cognitive and behavioral outcomes. Previous research showed that over one-third of mothers of children with disabilities have significant levels of depressive symptoms, a rate higher than the population at large. Infants and toddlers of depressed mothers have been shown to receive fewer intensive services and have been shown to interfere with uptake of EI services through impaired mother-child interactions. A preliminary study by the investigators found that over a third of mothers of infants and toddlers enrolled in EI in a large North Carolina county had severe depressive symptoms and depression histories. Fortunately, the investigators also found that when depressed mothers were provided with concrete, attainable skills for improving interactions with their child, the impact of depression on both mother and child was substantially reduced. Focusing on a depressed mother's child-centered speech and reciprocal communication also improves child outcomes, even when the child is cognitively compromised. However, none of these specialized services are part of EI best practices. Thus, EI is an ideal setting in which to integrate screening, referral and targeted skills for depressed mothers in order to improve parent-child interactions and ultimately, child outcomes.

This project will develop an intervention focused on communication between infants and toddlers with diagnosed or suspected developmental disabilities and their mothers who have depressive symptoms. The primary aim of the study is to test the feasibility and initial efficacy of embedding a language pedometer, the Language ENhancement Assessment/intervention system (LENA), into EI to teach mothers to increase child-centered speech and reciprocal communication, which have been linked to positive child outcomes, and to increase parenting efficacy in depressed mothers of children in EI.

While maternal depressive symptoms can disrupt developmentally stimulating, child-centered speech, simple tools to assess and provide feedback to mothers can improve the child-centered speech and reciprocal language interactions that positively impact child outcomes. Although the LENA has been used in other studies and shown improvements in mothers' child-centered speech, the system has not been used with mothers showing depressive symptoms or in the EI context. The investigators will examine the efficacy of using LENA in a pre-/post-intervention design. Specifically, the investigators will examine whether mothers' primarily independent use of the LENA with feedback has an impact on the child's language environment, parenting efficacy and maternal depressive symptoms.

The investigators will also conduct follow up data collection with participating mothers, which will be approximately 6 months after her last LENA recording. Follow up activities will involve having the mother conduct one more LENA recording and provide survey information over the phone, which will allow the investigators to determine residual effects of the study interventions, additional demographic information, and feedback for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older. Mothers who are 18 years can give consent independently.
* Be the biological or adoptive mother of an infant (6 weeks - 18 months old) or toddler (19 -32 months old) enrolled in EI at the time of recruitment; mothers must be the primary caretaker of the child.
* EI services are offered only to infants and toddlers up to the age of 36 months; this study caps the age of enrollment at 32 months to ensure that toddlers are continuously enrolled in EI during the data collection period.
* Able to independently give consent. Mothers must have adequate capacity to participate in the LENA intervention as well as understand what they will be asked to do as participants.
* Score 8 or higher on the Patient Health Questionnaire - (PHQ-9). This score is indicative of depressive symptoms.

Exclusion Criteria:

* Currently pregnant by self-report.
* Child is completely deaf

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2018-11-04 (Actual); Study Completion 2018-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Beeber, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Anne Wheeler, PhD, Principal Investigator — RTI International; Doré LaForett, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Durham Children's Developmental Services Agency, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Interest letters describing the study were mailed from the Part C research partner to mothers in April -June 2018. Interested mothers contacted the research team by phone or email, and were then screened for eligibility. Eligible mothers completed consent forms at their homes with researchers during the Baseline visit.
Groups:
- LENA With Feedback: Mothers who will run the Language ENhancement Assessment/intervention system with their young children, and will receive initial feedback from researchers on LENA output and how to enhance the home language environment.
  Language ENhancement Assessment/intervention system: The LENA with Feedback intervention will involve mothers running the Language ENhancement Assessment/intervention system, an audiorecorder language pedometer that records adult speech centered on the child, child vocalizations, and parent-child reciprocal turn-taking conversations. Researchers will provide an initial feedback session to mothers, which will include reviewing the LENA visual output from the previous recording and how mothers can access the output on their own for future recordings. Mothers will independently use the LENA system and access the output on their own.
Period: Overall Study
Arm/Group | LENA With Feedback
Started | 10
Time 1 Data Collection (T1) | 10
LENA Baseline | 10
LENA Time 1 | 10
LENA Time 2 | 10
LENA Time 3 | 10
LENA Time 4 | 9
LENA Time 5 | 8
Time 2 Data Collection (T2) | 8
Completed | 8
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | LENA With Feedback
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (5.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10
LENA Adult Word Count - Number of Words [Mean (Standard Deviation); unit: number of words] — The Language Enhancement/Intervention System (LENA), which records adult-child vocalizations, measures the number of the target adult's (e.g., parent) child-directed words (child-directed speech). The total possible range is 0-n, where higher scores indicate an increased number of child-directed words spoken by the target adult and higher degrees of a language-rich environment. Lower scores indicate fewer words spoken by the target adult and represent an environment that is not language-rich.
  number of words | 12274.20 (6142.03)
Parenting Sense of Competence [Mean (Standard Deviation); unit: units on a scale] — The Parenting Sense of Competence Scale is a 17-item measure assessing parental competence. Each item is rated on a 6 point Likert scale anchored by 1 = "Strongly Disagree" and 6 = "Strongly Agree". The Efficacy subscale measures feelings of efficacy as a parent. It has 7 questions (1,6,7,10,11,13,15), producing a range of 6-42. Higher scores indicate greater self-efficacy. Lower scores mean more impairment.
  units on a scale | 17.90 (7.94)
Patient Health Questionnaire - 9 [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionnaire - 9 (PHQ-9) is a depression scale used to assess brief depression severity by rating symptoms and functional impairment experienced in the last two weeks. Nine questions are scored on a range from 0-3; "0" = not at all, "1" =several days, "2" = more than half the days, and "3" = nearly every day. The total possible range is 0-27, with higher scores indicating more depressive symptoms (0-4 = minimal depression, 5-9 = mild depression, 10-14 = moderate depression, 15-19 = moderately severe depression, and 20-27 = severe depression).
  units on a scale | 4.8 (6.05)
LENA Mother/Child Turn Taking [Mean (Standard Deviation); unit: number of turns] — The LENA system, which records adult-child vocalizations, measures the number of conversational turns between the target adult (e.g., parent) and child. The total possible range is 0-n, where higher scores indicate an increased number of turns (back-and-forth, or "reciprocal" language exchanges) between the adult and child, reflecting higher degrees of a language-rich environment. Lower scores indicate fewer conversational turns between the adult and child, and represent an environment that is not language-rich.
  number of turns | 416.7 (257.23)
LENA Child Vocalization [Mean (Standard Deviation); unit: number of vocalizations] — The LENA system, which records adult-child vocalizations, measures the number of vocalizations of the target child. The total possible range is 0-n, where higher scores indicate an increased number of vocalizations from the child, reflecting higher levels of language development. Lower scores indicate fewer vocalizations from child, and represent lower levels of language development.
  number of vocalizations | 1726.00 (651.35)
Generalized Anxiety Disorder - 7 [Mean (Standard Deviation); unit: units on a scale] — The Generalized Anxiety Disorder 7-item (GAD-7) is a self-report screening of anxiety symptoms examining frequency the of specific behaviors within the last two-weeks (e.g., not at all - nearly every day). A total score is calculated and compared to pre-determined cutoffs to help guide professionals in next steps for evaluation and treatment. The GAD-7 consists of seven items which are scored from zero to three. Scores range from 0-21, with higher scores reflecting more severe anxiety symptoms. The cut-off scores for mild, moderate and severe anxiety symptoms are 5, 10 and 15 respectively.
  units on a scale | 4.20 (6.07)

OUTCOME MEASURES:

1. Primary Outcome: LENA Adult Word Count Score at 6 Weeks
Description: The Language Enhancement/Intervention System (LENA), which records adult-child vocalizations, measures the number of the target adult's (e.g., parent) child-directed words (child-directed speech). The total possible range is 0-n, where higher scores indicate an increased number of child-directed words spoken by the target adult and higher degrees of a language-rich environment. Lower scores indicate fewer words spoken by the target adult and represent an environment that is not language-rich.
Time Frame: at 6 weeks
Measure: Mean (Standard Deviation); unit: number of words
Arm/Group | LENA With Feedback
Number analyzed (Participants) | 8
number of words | 18391.25 (8500.97)

2. Secondary Outcome: Parenting Sense of Competence Scale Efficacy Subscale Score at 6 Weeks
Description: The Parenting Sense of Competence Scale is a 17-item measure assessing parental competence. Each item is rated on a 6 point Likert scale anchored by 1 = "Strongly Disagree" and 6 = "Strongly Agree". The Efficacy subscale measures feelings of efficacy as a parent. It has 7 questions (1,6,7,10,11,13,15), producing a range of 6-42. Higher scores indicate greater self-efficacy. Lower scores mean more impairment.
Time Frame: at 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LENA With Feedback
Number analyzed (Participants) | 8
units on a scale | 19.00 (10.85)

3. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9) Score at 6 Weeks
Description: The Patient Health Questionnaire - 9 (PHQ-9) is a depression scale used to assess brief depression severity by rating symptoms and functional impairment experienced in the last two weeks. Nine questions are scored on a range from 0-3; "0" = not at all, "1" =several days, "2" = more than half the days, and "3" = nearly every day. The total possible range is 0-27, with higher scores indicating more depressive symptoms (0-4 = minimal depression, 5-9 = mild depression, 10-14 = moderate depression, 15-19 = moderately severe depression, and 20-27 = severe depression).
Time Frame: at 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LENA With Feedback
Number analyzed (Participants) | 8
units on a scale | 4.25 (4.06)

4. Secondary Outcome: LENA Mother/Child Turn-Taking Score at 6 Weeks
Description: The LENA system, which records adult-child vocalizations, measures the number of conversational turns between the target adult (e.g., parent) and child. The total possible range is 0-n, where higher scores indicate an increased number of turns (back-and-forth, or "reciprocal" language exchanges) between the adult and child, reflecting higher degrees of a language-rich environment. Lower scores indicate fewer conversational turns between the adult and child, and represent an environment that is not language-rich.
Time Frame: at 6 weeks
Measure: Mean (Standard Deviation); unit: number of turns
Arm/Group | LENA With Feedback
Number analyzed (Participants) | 8
number of turns | 365.38 (259.00)

5. Secondary Outcome: LENA Child Vocalization Score at 6 Weeks
Description: The LENA system, which records adult-child vocalizations, measures the number of vocalizations of the target child. The total possible range is 0-n, where higher scores indicate an increased number of vocalizations from the child, reflecting higher levels of language development. Lower scores indicate fewer vocalizations from child, and represent lower levels of language development.
Time Frame: at 6 weeks
Measure: Mean (Standard Deviation); unit: number of vocalizations
Arm/Group | LENA With Feedback
Number analyzed (Participants) | 8
number of vocalizations | 1199.13 (759.47)

6. Secondary Outcome: Generalized Anxiety Disorder (7-Item) Score at 6 Weeks
Description: The Generalized Anxiety Disorder 7-item (GAD-7) is a self-report screening of anxiety symptoms examining frequency the of specific behaviors within the last two-weeks (e.g., not at all - nearly every day). A total score is calculated and compared to pre-determined cutoffs to help guide professionals in next steps for evaluation and treatment.The GAD-7 consists of seven items which are scored from zero to three. Scores range from 0-21, with higher scores reflecting more severe anxiety symptoms. The cut-off scores for mild, moderate and severe anxiety symptoms are 5, 10 and 15 respectively.
Time Frame: at 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LENA With Feedback
Number analyzed (Participants) | 8
units on a scale | 3.63 (4.37)

ADVERSE EVENTS:
Time Frame: Beginning at screening call and up to 6 months after T2 data collection (e.g., an average of 1 year)
Arm/Group | LENA With Feedback
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-12): https://cdn.clinicaltrials.gov/large-docs/41/NCT03480841/Prot_SAP_001.pdf